CLINICAL TRIAL: NCT02522507
Title: A Peer E-mentoring Intervention to Improve Transition to Employment for Youth With Physical Disabilities
Brief Title: A Peer E-mentoring Intervention to Improve Employment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Ability Online (Other); University of Toronto (Other); The Hospital for Sick Children (Other); University of Ottawa (Other); Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 15-590
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy; Spina Bifida; Juvenile Arthritis; Spinal Cord Injury; Muscular Dystrophy; Physical Disability
MeSH Terms: conditions — Cerebral Palsy; Spinal Dysraphism; Arthritis, Juvenile; Spinal Cord Injuries; Muscular Dystrophies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empowering youth towards employment (Experimental): This is a behavioural e-mentor intervention. Trained mentors will facilitate employment readiness learning and engage youth in discussions over a 12-week period. Each week the mentors will introduce a new employment topic and will engage youth in a discussion and answer questions.
  Interventions: Behavioral: Empowering youth towards employment
- Control group (No Intervention): The control group will have access to the employment activities during the 12-week employment readiness learning but will not have access to a mentor.

INTERVENTIONS:
Behavioral: Empowering youth towards employment — Experimental: Empowering youth towards employment This is a behavioural e-mentor intervention. Trained mentors will facilitate employment readiness learning and engage youth in discussions over a 12-week period. Each week the mentors will introduce a new employment topic and will engage youth in a discussion and answer questions.
  Arms: Empowering youth towards employment

SUMMARY:
Despite the strong business case of hiring people with disabilities, a significant proportion of youth with disabilities leave high school and neither work nor continue their education and are unprepared to meet the demands of a work environment. Although youth with disabilities have much to gain from employment readiness programs, they are often excluded from, or have limited access to school and community vocational programs. One encouraging approach to address gaps in vocational programming is through peer mentoring, which may facilitate a smoother transition to adulthood by offering support to enhance coping skills. Despite the increase in online communities, little is known about their impact on vocational mentoring for youth with physical disabilities and their parents. The purpose of this study is to develop, implement and assess the feasibility of an online peer mentor employment readiness intervention for youth with physical disabilities and their parents to improve their self-efficacy, career maturity and social support.

DETAILED DESCRIPTION:
Our primary OBJECTIVE is: (1) to develop, implement and assess the feasibility of an online peer mentor employment readiness intervention for youth with physical disabilities and their parents to improve their self-efficacy, career maturity and social support.

A mixed methods feasibility randomized controlled trial design will be conducted to develop and assess the usability of "Empowering youth towards Employment" intervention. Youth (aged 15-25) with physical disabilities and their parents will be randomly assigned to a control or experimental group (12-week, interactive intervention, moderated by peer mentors). A qualitative thematic analysis will be conducted to analyze the content of discussion forums. Interviews with youth, parents and mentors will also be conducted about their experiences in the intervention.

ELIGIBILITY:
Inclusion criteria for youth participants:

* Able to read/write in English;
* A diagnosed physical disability (i.e., cerebral palsy, muscular dystrophy, spinal cord injury etc.); (4) currently enrolled in or have completed a high school diploma in the applied / academic stream (to screen for cognitive impairment);
* Aged 15-25;
* Have access to a computer and internet;
* Have no paid work experience.

Inclusion criteria for Parents:

* Are the parent of a youth meeting above inclusion criteria
* Can read/write in English
* Have access to a computer with Internet

Exclusion Criteria:

* Recently completed or currently participating in another employment readiness or peer support intervention.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change in career maturity inventory--attitude scale (CMI-AS) | baseline (1-week pre-study arm 1), 12 weeks (post-study arm 1)

SECONDARY OUTCOMES:
Change in family empowerment scale | baseline (1-week pre-study arm 1), 12 weeks (post-study arm 1)
Change in multi-dimensional scale of perceived social support | baseline (1-week pre-study arm 1), 12 weeks (post-study arm 1)
Change in Arc's self-determination scale | baseline (1-week pre-study arm 1), 12 weeks (post-study arm 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lindsay S, Cagliostro E, Leck J, Stinson J. A 12-Week Electronic Mentoring Employment Preparation Intervention for Youth With Physical Disabilities: Pilot Feasibility Randomized Controlled Trial. JMIR Pediatr Parent. 2019 Mar 29;2(1):e12088. doi: 10.2196/12088. PMID 31518315
- [Derived] Lindsay S, Cagliostro E, Stinson J, Leck J. A 4-Week Electronic-Mentoring Employment Intervention for Youth With Physical Disabilities: Pilot Randomized Controlled Trial. JMIR Pediatr Parent. 2019 Apr 24;2(1):e12653. doi: 10.2196/12653. PMID 31518302
- [Derived] Lindsay S, Stinson J, Stergiou-Kita M, Leck J. Improving Transition to Employment for Youth With Physical Disabilities: Protocol for a Peer Electronic Mentoring Intervention. JMIR Res Protoc. 2017 Nov 16;6(11):e215. doi: 10.2196/resprot.8034. PMID 29146566